CLINICAL TRIAL: NCT07247097
Title: ELDORADO: a Randomized Phase II Trial of Elranatamab or Daratumumab in Combination With Lenalidomide, Bortezomib, and Dexamethasone (RVd Lite) in Newly Diagnosed, Transplant Ineligible/Deferred Multiple Myeloma
Brief Title: ELDORADO: Elranatamab Versus Daratumumab in Combination With RVd Lite for Newly Diagnosed Transplant Ineligible/Deferred Multiple Myeloma
Acronym: ELDORADO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-699
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Newly Diagnosed Multiple Myeloma; Transplant Ineligible; Newly Diagnosed Multiple Myeloma (NDMM)
Keywords: NDMM; multiple myeloma; ELDORADO; RVd lite; transplant ineligible/deferred
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Bortezomib; Injections; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elranatamab with lenalidomide, bortezomib, and dexamethasone (elra-RVd lite) (Experimental): The first 10 patients will enroll in the elranatamab arm for a one 14-day safety run-in cycle. Elranatamab and dexamethasone will be administered at pre-determined doses on days 1, 4, and 8 of the cycle. After randomization occurs, patients in the elra-RVd lite arm will complete 24 cycles (each cycle is 28 days) of treatment. On day 1 of each cycle and day 15 of cycle 1, the pre-determined dose of elranatamab will be administered via subcutaneous injection. On days 1-21 of each cycle, patients will take the pre-determined dose of oral lenalidomide. One days 1, 8, and 15 of cycles 1-8, the pre-determined dose of bortezomib will be administered via subcutaneous injection. After completion of 24 treatment cycles, patients who have had two MRD negative tests, one year apart, may discontinue treatment and enter the observation phase of the trial. Patients who have not had two MRD negative tests one year apart, may continue elranatamab lenalidomide treatment for another 24 cycles.
  Interventions: Drug: Elranatamab (PF-06863135); Drug: Lenalidomide; Drug: Bortezomib for Injection; Drug: Dexamethasone
- Daratumumab with lenalidomide, bortezomib, and dexamethasone (dara-RVd lite) (Experimental): After randomization occurs, patients in the dara-RVd lite arm will complete 24 cycles (each cycle is 28 days) of treatment. On days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7+, the pre-determined dose of daratumumab will be administered via subcutaneous injection. On days 1-21 of each cycle, patients will take the pre-determined dose of oral lenalidomide. One days 1, 8, and 15 of cycles 1-8, the pre-determined dose of bortezomib will be administered via subcutaneous injection. On days 1, 2, 8, 9, 15, 16 of cycles 3+, as well as days 22 and 23 of cycles 1 and 2, patients will take the pre-determined dose of oral dexamethasone.
  Interventions: Drug: Daratumumab and Hyaluronidase-fihj; Drug: Lenalidomide; Drug: Bortezomib for Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elranatamab (PF-06863135) — Elranatamab is a bispecific IgG2 kappa monoclonal antibody.
  Arms: Elranatamab with lenalidomide, bortezomib, and dexamethasone (elra-RVd lite)
Drug: Daratumumab and Hyaluronidase-fihj — Daratumumab is an immunoglobulin G1 kappa human monoclonal antibody against CD38 antigen.
  Arms: Daratumumab with lenalidomide, bortezomib, and dexamethasone (dara-RVd lite)
Drug: Lenalidomide — Lenalidomide is a thalidomide analogue and an immunomodulatory agent with antiangiogenic properties.
Drug: Bortezomib for Injection — Bortezomib for injection is a small molecule proteosome inhibitor.
Drug: Dexamethasone — Dexamethasone is a synthetic adrenocortical steroid.

SUMMARY:
This research study is being done to compare the efficacy and safety of the combination of elranatamab, lenalidomide, bortezomib, dexamethasone versus the combination of daratumumab, lenalidomide, bortezomib, dexamethasone for patients with newly diagnosed, transplant ineligible/deferred multiple myeloma.

DETAILED DESCRIPTION:
The ELDORADO trial is a phase 2, randomized, open label, multicenter study that will enroll approximately 160 patients (10 patient safety run and 150 patients for randomization) to compare the efficacy and safety of the combination of elranatamab, lenalidomide, bortezomib, dexamethasone versus the standard combination of daratumumab and hyaluronidase, lenalidomide, bortezomib, dexamethasone in newly diagnosed, transplant ineligible/deferred multiple myeloma patients. Pfizer, Inc. is supporting this research by providing the study drug, elranatamab, and funding for research activities. Patients will receive treatment for 24 cycles. For patients who meet certain testing parameters, some patients may be able to discontinue treatment and be observed. Other patients may continue with the treatment that they have been receiving until disease progression. Patients may discontinue treatment if they experience unacceptable adverse events, their condition changes rendering them unacceptable for further treatment, they experience intercurrent illness that prevents further administration of treatment, they demonstrate an inability or unwillingness to comply with the medication regimen and/or documentation requirements, or they withdraw from the study. Patients will be followed for a period of 5 years from when the last participant discontinues treatment. The majority of this follow up will not be in person and will be through review of the patients' charts. The U.S. FDA has not approved the combination of elranatamab or daratumumab with lenalidomide, bortezomib, and dexamethasone (elra-RVd lite or dara-RVd lite) as a treatment for any disease. Elranatamab is a bispecific antibody, meaning it can attach to two different things at the same time. Elranatamab, specifically, connects to cancer cells, as well as to a certain type of immune cells, called T cells, to help the immune system attack and destroy the cancer cells. Daratumumab recognizes and attaches to a protein found on the surface of cancer cells, called CD38. This aids the immune system in identifying and destroying cancer cells. Lenalidomide is an immunomodulatory drug. Immunomodulatory drugs help control or adjust how the immune system works, whether it is too weak or too aggressive to more effectively fight infections and cancers. Bortezomib is a proteasome inhibitor, meaning it blocks proteasome in cells. Proteasome aids in cell growth and development. When proteasome is blocked, damaged proteins build up, stressing a cancer cell, and eventually cause cell death. Dexamethasone is a glucocorticoid (a substance that stops inflammation caused by immune system disorders) that has shown significant activity in myeloma. It is believed to aid in anti-myeloma effects, which may lead to the destruction of myeloma cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Newly diagnosed multiple myeloma, with monoclonal plasma cells in the bone marrow ≥10% or a biopsy proven plasmacytoma and either CRAB criteria or biomarker of malignancy

  a. CRAB criteria, one or more of the following: i. Hypercalcemia: serum calcium (>1 mg/dL) higher than the upper limit of normal or >11 mg/dL ii. Renal insufficiency: creatinine clearance <40 mL/min (calculated per local practice) or serum creatinine >2 mg/dL iii. Anemia: hemoglobin value >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL iv. Bone lesions: one or more lytic lesions on skeletal radiography, CT, or PET CT b. Biomarker of malignancy (one or more of the following): i. Clonal bone marrow plasma cells ≥60% ii. Involved:uninvolved serum free light chain ratio ≥100 iii. >1 focal lesion on magnetic resonance imaging (MRI)
* Measurable disease as defined by one of the following:

  1. Serum monoclonal protein ≥0.5 g/dL. For IgA monoclonal protein, total IgA >500 mg/dL is allowable.
  2. Urine monoclonal protein ≥200 mg/24 hours
  3. Involved serum free light chain ≥100 mg/L with abnormal free light chain ratio
* Not considered eligible for high dose melphalan and autologous stem cell transplant per treating investigator or plan for deferred high dose melphalan and autologous stem transplant
* ECOG performance status of 0-2
* ANC ≥1000/μL. G-CSF is not permitted within 14 days of screening.
* Platelet count ≥75,000/µL. Platelet count ≥50,000/µL is permitted if bone marrow is >50% involved. Platelet transfusion and thrombopoietin receptor agonists are not permitted within 7 days of screening.
* Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
* Calculated creatinine clearance of ≥ 30 mL/min, not requiring dialysis, with calculation per local practice.
* Serum bilirubin values < 1.5 x ULN. Isolated bilirubin x 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (e.g. total bilirubin <3 mg/dL and normal direct bilirubin); and
* Serum aspartate transaminase (ALT) and aspartate transaminase (AST) values < 2.5 × the upper limit of normal (ULN) of the institutional laboratory reference range.
* Must be able to comply with thromboembolism prophylaxis with e.g. acetylsalicylic acid (ASA), apixaban, rivaroxaban, lower molecular weight heparin, or equivalent.
* Females of childbearing potential (FCBP) must:

  1. Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy within 10-14 days, with the second test within 24 hours of starting lenalidomide. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
  2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use and be able to comply with two reliable forms of contraception as defined by lenalidomide Risk Evaluation and Mitigation Strategy (REMS) program.
* Male subjects must follow the lenalidomide REMS.
* Ability and the willingness to undergo repeat bone marrow biopsy assessments.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior or current systemic therapy for any plasma cell disorder. An exception is emergency use of corticosteroids (equivalent to dexamethasone 40 mg daily for four days). After discussion with the principal investigator. one cycle of standard of care myeloma therapy (without anti-CD38 monoclonal antibody) is permissible to allow for stabilization of disease, during screening/prior to enrollment.
* Pregnancy, currently breastfeeding, or planned breastfeeding.
* Participant plans to father a child while enrolled in the study or within 100 days after last dose of study treatment.
* Prior history of malignancies, other than MM, unless the patient has completed definitive treatment and has been free of the disease for ≥3 years. Patients who are free of disease <3 years may enroll after approval of the PI (e.g. localized breast cancer considered to have very low risk of recurrence). Exceptions include the following (i.e. the following are eligible to participate):

  1. Basal or squamous cell carcinoma of the skin
  2. Carcinoma in situ of the cervix
  3. Ductal carcinoma in situ of the breast
  4. Incidental histologic finding of prostate cancer (T1a or T1b) managed with surveillance
  5. Other malignancies of clinically localized disease may be permitted to enroll after discussion with the Sponsor-Investigator
* Patients with plasma cell leukemia at time of screening, POEMS syndrome, or primary AL amyloidosis are excluded from this trial.
* Seropositive for HIV infection.
* Hepatitis B viral load positive.
* Hepatitis C viral load positive.
* Peripheral neuropathy ≥grade 2.
* Patient has a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to:

  1. Congestive heart failure (New York Heart Association [NYHA] Class 3 or 4)
  2. Unstable angina
  3. Clinically significant, uncontrolled cardiac arrhythmia such a 2nd degree or 3rd degree atrioventricular block
  4. Recent (within the preceding 6 months) myocardial infarction or stroke
  5. Severe non-ischemic cardiomyopathy.
  6. Uncontrolled hypertension
  7. Diabetes mellitus with >2 episodes of ketoacidosis in the preceding 12 months
  8. Chronic obstructive pulmonary disease (COPD) requiring >2 hospitalizations in the preceding 12 months.
  9. Acute diffuse infiltrative pulmonary disease.
  10. Active bacterial, viral, or fungal infection
  11. Stroke, transient ischemic attack, or seizure within six months of starting treatment.
* Patient has any other medical, psychiatric, or social condition that would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results.
* Major surgery within 4 weeks prior to C1D1. Kyphoplasty or vertebroplasty are not considered major surgery.
* Received an investigational drug (or vaccine) or used an invasive investigational medical device within four weeks before screening or is currently enrolled in an interventional investigational study.
* Live or live-attenuated vaccine within 30 days prior to C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion Patients who test Negative for Minimal Residual Disease (MRD) at 10^-5 after 4 Treatment Cycles | Day 1 of Cycle 1 (each cycle is 28 days) to Day 28 of Cycle 4.
  Evaluated at 1 x 10^-5 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who test negative for MRD at 10^-5 after 4 treatment cycles will be compared between the elran-RVd lite arm and the dara-RVd lite arm.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Day 1 of Cycle 1 (each cycle is 28 days) to documentation of disease progression or death from any cause (up to 5 years). Patients who have not progressed or died are censored at the date last known progression-free.
  Progression-free survival (PFS) is the time from randomization to disease progression or death from any cause. PFS distributions will be calculated using the Kaplan-Meier method. PFS will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Overall Survival (OS) | Day 1 of Cycle 1 (each cycle is 28 days) to documentation of death due to any cause or censored at the date last known alive, up to 5 years from study registration.
  Overall survival (OS) is the time from start of treatment to death due to any cause. OS distributions will be calculated using the Kaplan-Meier method. OS will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Overall Response Rate (ORR) | Day of initiation of first response to the first documentation of disease progression or death, up to 5 years after registration. Patients who have not progressed or died are censored at the date last known progression-free.
  Overall response rate (ORR) is the proportion of patients achieving partial response or better, along with very good partial response and complete response per the International Myeloma Working Group Response Criteria (IMWG). All IMWG response categories will require one confirmation. ORR will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Proportion Patients who test Negative for Minimal Residual Disease (MRD) at 10^-5 after 12 Treatment Cycles | Day 1 of Cycle 1 (each cycle is 28 days) to Day 28 of Cycle 12.
  Evaluated at 1 x 10^-5 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who test negative for MRD at 10^-5 after 12 treatment cycles will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Proportion Patients who test Negative for Minimal Residual Disease (MRD) at 10^-6 after 4 Treatment Cycles | Day 1 of Cycle 1 (each cycle is 28 days) to Day 28 of Cycle 4.
  Evaluated at 1 x 10^-6 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who test negative for MRD at 10^-6 after 4 treatment cycles will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Proportion Patients who Remain Negative for Minimal Residual Disease (MRD) at 10^-5 for 12 Months | Day of first negative MRD test to study completion (up to 5 years).
  12-month sustained MRD is defined as two MRD negative results a minimum of 12 months apart (with a window of four weeks). Evaluated at 1 x 10^-5 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who remain negative for MRD at 10^-5 for 12 months will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Proportion Patients who Remain Negative for Minimal Residual Disease (MRD) at 10^-6 for 12 Months | Day of first negative MRD test to study completion (up to 5 years).
  12-month sustained MRD is defined as two MRD negative results a minimum of 12 months apart (with a window of four weeks). Evaluated at 1 x 10^-6 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who remain negative for MRD at 10^-6 for 12 months will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Proportion Patients who test Negative for Minimal Residual Disease (MRD) at 10^-6 after 12 Treatment Cycles | Day 1 of Cycle 1 (each cycle is 28 days) to Day 28 of Cycle 12.
  Evaluated at 1 x 10^-6 using next generation sequencing (NGS) to detect clonal sequences. The proportions will be compared using the Cochran-Mantzel-Haenszel test, stratified by the randomization stratification factors. A one-sided significance level of 0.05 will be used. Patients without successful baseline minimal residual disease (MRD) testing will not be evaluated for MRD response. Proportion patients who test negative for MRD at 10^-6 after 12 treatment cycles will be compared between the elran-RVd lite arm and the dara-RVd lite arm.
Depth of Response using Peripheral Blood Mass Spectrometry | Day 1 of cycle 1 (each cycle is 28 days) to day 28 of cycle 24.
  For the first 50 patients (including the safety run in patients), peripheral blood will be collected for monoclonal protein measurement by mass spectrometry. Mass spectrometry to measure serum monoclonal protein as a form of peripheral blood minimal residual disease (MRD) determination will be compared to the performance of an established assay for measuring minimal residual disease in the bone marrow using next generation sequencing (NGS) by Clonoseq at 10^-5 threshold. The study will use spectrometry with a clonotypic-based approach using the M-Insight assay.
Number of Patients who Experience Adverse Events (AEs) | Day 1 of cycle 1 (each cycle is 28 days) to day 28 of the patient's last treatment cycle (up to 48 cycles).
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Assessment for cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) using the American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Attribution of the adverse event (AE) will be determined as definite (clearly related to the study treatment), probably (likely related to the study treatment), possible (may be related to the study treatment), unlikely (doubtfully related to the study treatment), or unrelated (clearly not related to the study treatment). A "serious" adverse event is a regulatory definition and is based on subject or event outcome or action criteria usually associated with events that post a threat to a subject's life or functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Dr. Andrew Yee at 617-724-4000. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation